CLINICAL TRIAL: NCT01776073
Title: Evaluation of a Patient Navigation System to Reduce Time to Waitlisting for Potential Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rachel Patzer, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00060661; Mason-01 (Other: Other)
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: End-Stage Renal Disease
Keywords: Transplantation; Healthcare Disparities; Quality Assurance
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient navigation (Experimental): In addition to receiving the standard of care, these patients will be connected with a patient navigator who will provide personalized assistance with regard to completion of the pre-waitlisting process
  Interventions: Behavioral: Patient Navigation
- Standard of Care (No Intervention): These patients will receive the standard of care, which includes assistance from the current Emory Transplant Center team of social workers, physicians, and other support staff with regard to completion of the pre-waitlisting process

INTERVENTIONS:
Behavioral: Patient Navigation
  Arms: Patient navigation

SUMMARY:
The purpose of this study is to measure the effect of introducing a patient navigator to guide high and moderate risk patients through the pre-waitlisting phases of the kidney transplant process. Patients identified as being at high and moderate risk of delay to waitlisting will be linked with a patient navigator, who will facilitate their completion of pre-waitlisting requirements. We believe that patients who are randomized to a patient navigator will be more likely to complete the pre-waitlisting process and will complete the process more quickly than high and moderate risk patients who do not receive additional assistance from a patient navigator.

DETAILED DESCRIPTION:
The investigators plan to implement a newly developed risk assessment tool that uses medical and demographic indicators to estimate the probability of waitlisting for all patients beginning the transplant process at the Emory Transplant Center. Medical secretaries will collect information about patients' medical and demographic characteristics during the appointment scheduling phone call. This information will be entered into the REDCap risk assessment tool, which will be used to calculate the probability of waitlisting. A previously defined cut-off will be used to categorize the risk of delay to waitlisting.

A random subset of patients identified as being at high and moderate risk of delay to waitlisting will be connected with a patient navigator, who will be available not only to answer questions, but also to manage clinical information prior to, during, and following transplantation. The navigator will work to identify potential barriers and to ensure that the most up-to-date clinical information has garnered responses at the nurse and physician levels.

The effect of connecting high and moderate risk patients with a patient navigator on time to waitlisting and rate of waitlisting will be analyzed to determine whether such a program is an effective means of increasing access to transplant for patients who are likely to face financial, racial, and demographic barriers.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant candidates older than 18 years of age at Emory Transplant Center

Exclusion Criteria:

* There are no exclusion criteria that would limit subject participation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2013-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Time from evaluation to waitlisting in referred patients; Rate of pre-transplant evaluation completion | 1 year

SECONDARY OUTCOMES:
Time from referral to evaluation appointment | 1 year
Time from referral to initial listing (active or inactive) | 1 year
Time from referral to transplant | 1 year

OTHER OUTCOMES:
Rate of loss to follow-up; Rate of failure to show for evaluation appointment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Patzer, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States